CLINICAL TRIAL: NCT06556901
Title: Evaluation of the Feeling of General Practitioners in the Management of Patients Who Claim to be Electrosensitive
Brief Title: Management of Patients Who Claim to be Electrosensitive
Acronym: IEI CEM EN MED
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0155
Record Dates: First submitted 2021-06-04; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Electromagnetic Field
Keywords: qualitative study; environmental exposure
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective study about reasons for consultations — retrospective study about reasons for consultations

SUMMARY:
Know qualitatively the ways to deal with these patients, in general medicine in Brittany, and the difficulties encountered, through thematic and lexicometric analysis of responses

DETAILED DESCRIPTION:
The Ministry of Health instructed the French society of medicine work (Dr Pougnet for the Brest CHRU) to coordinate the drafting of practical guides for the management of people claiming to have IEI-CEM (Intolerance Environmental Idiopathic in the Fields ElectroMagnetic) for care physicians primary (general practitioners). To meet this mission, it is necessary to know qualitatively the difficulties encountered by general practitioners during the management of these people.

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria will be to be general practitioners, to have practiced between 01/01/2018 and 12/31/2018.

Exclusion Criteria:

* be other practionners

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population of general practitioners practicing in Brittany in 2018. Population assessed by the ODM between 3000 and 3200 liberal general practitioners
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
principal | 2 years
  The main endpoint is to have taken care of a patient who claims to have electromagnetic sensibility.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanderstraeten J, Verschaeve L. Biological effects of radiofrequency fields: Testing a paradigm shift in dosimetry. Environ Res. 2020 May;184:109387. doi: 10.1016/j.envres.2020.109387. Epub 2020 Mar 12. PMID 32182484